CLINICAL TRIAL: NCT06464029
Title: Pathways Mediating Impaired Postural Control in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUR-2023-31981
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: 40 healthy older adults and 40 young adults. Potential volunteers for the study will be recruited from a list of volunteers at the University of Minnesota or study information pamphlets distributed people who express an interest in participating (e.g. at research events, support group meetings, or to colleagues of participants tested). Interested individuals will self-identify and contact our research staff for further information.
- Experimental: 40 people with Parkinson's disease. Potential volunteers will be recruited from the Movement Disorders Clinic at the University of Minnesota Medical Center. Patients that are referred to this center for standard-of-care evaluations will be seen by a movement disorders neurologist. Patients will be evaluated as per standard of care, regardless of whether they are interested in participating in research protocols.

SUMMARY:
The purpose of this project is to use transcranial magnetic stimulation (TMS) to explore the state of excitability of corticocortical and corticofugal (cortex to spinal cord, cortex to brainstem to spinal cord) pathways that project to muscles that control the legs and trunk in people with Parkinson's disease. The outcome variables will be further analyzed to understand their relationship to quantitative measures of postural instability and gait dysfunction. As such, the project can be classified as basic physiologic research. The protocol is not designed to determine if measures of corticocortical or corticofugal excitability can be used as a biomarker to predict disease progression.

ELIGIBILITY:
Inclusion Criteria:

Participants with Parkinson's disease

* Diagnosis of idiopathic PD or dystonia as determined by a movement disorders neurologist in accordance with the UK Society Brain Bank diagnostic criteria.
* Age 45-80 years.
* Able to ambulate independently without the use of an assistive device (e.g. cane) for 50 meters.

Healthy Older Adults (Control participants)

* Age 45-80 years (this group will be age and sex-matched to the PD group)
* Able to ambulate independently without the use of an assistive device (cane or walker)

Healthy Young Adults

* Age 21-44 years (this group will be age and sex-matched to the PD group)
* Able to ambulate independently without the use of an assistive device (cane or walker)

Exclusion Criteria:

* Subjects who describe a history of a frequent vasovagal syncope (fainting) in response to blood, emotional stress, or sensory triggers.
* Subjects who are on anti-coagulant medications.
* Any musculoskeletal disorder that affects the ability to stand.
* History of seizures, epilepsy, stroke, multiple sclerosis, or traumatic brain injury.
* Intracranial metallic or magnetic devices.
* Pacemaker or any implanted device.
* History of surgery on blood vessels, brain or heart.
* Unexplained, recurring headaches or concussion within the last six months.
* Moderate to severe hearing impairment.
* Subjects who are pregnant.
* Dementia diagnosis
* Other significant neurological disorders that may affect participation or performance in the study
* Implanted deep brain stimulator or other neurosurgeries to treat PD.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with PD will undergo an initial screening for inclusion/exclusion criteria by their clinician based on findings obtained during their routine clinical appointment.
  Potential control participants will be screened for inclusion/exclusion criteria during an initial phone call.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
average gate speed | baseline
  Participants will walk on an overground pressure walkway (GAITRite, Franklin, NJ) that provides spatiotemporal measures of walking. In addition, they will wear a set of wearable sensors (APDM Inc., Opals) attached to the feet, wrists and trunk (lumbar and sternum) to capture whole-body motion.
stride length | baseline
  Participants will walk on an overground pressure walkway (GAITRite, Franklin, NJ) that provides spatiotemporal measures of walking. In addition, they will wear a set of wearable sensors (APDM Inc., Opals) attached to the feet, wrists and trunk (lumbar and sternum) to capture whole-body motion.
cadence | baseline
  Participants will walk on an overground pressure walkway (GAITRite, Franklin, NJ) that provides spatiotemporal measures of walking. In addition, they will wear a set of wearable sensors (APDM Inc., Opals) attached to the feet, wrists and trunk (lumbar and sternum) to capture whole-body motion.
turn speed | baseline
  Participants will walk on an overground pressure walkway (GAITRite, Franklin, NJ) that provides spatiotemporal measures of walking. In addition, they will wear a set of wearable sensors (APDM Inc., Opals) attached to the feet, wrists and trunk (lumbar and sternum) to capture whole-body motion.
ankle rigidity | 25mins
  Quantitative measures of rigidity will be obtained using a custom-built robotic manipulandum. The manipulandum moves the ankle through a sinusoidal or triangular range of motion (25 deg of plantar flexion to 5 degrees of dorsiflexion; modified as needed for participant's range of motion) while measuring the resistive torque generated by ankle impedance.
Root mean square of the excursion of the center of pressure | 5mins
  Participants will stand on a set of force platforms that measures the forces and pressures beneath the feet. Primary outcome
single pulse TMS | 1.5hrs
  A measure of the excitability of corticospinal pathways. Primary outcome variables: Peak-to-peak amplitude of the motor evoked potential (MEP) responses to TMS in lower limb and trunk muscles.
Paired-Pulse TMS (Intracortical excitability): | 1hr
  A measure of the excitability of intracortical (motor cortex-motor cortex) inhibitory (short-intracortical inhibition, SICI) and excitatory (short-intracortical inhibition, ICF) networks.
  Primary outcome variables: Peak-to-peak amplitude of the motor evoked potential (MEP) responses to TMS in lower limb and trunk muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Colum MacKinnon, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States